CLINICAL TRIAL: NCT07183137
Title: A Prospective Observational Study on Metabolic Surgery for the Treatment of Metabolic Syndrome
Brief Title: Metabolic Surgery for Metabolic Syndrome
Status: Completed | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-S008
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Syndrome (MetS); Hypertension (HTN); Obesity; T2; T2DM; Bariatric Surgery; Metabolic Surgery
Keywords: bariatric surgery; blood pressure; hypertension; T2DM; obesity
MeSH Terms: conditions — Metabolic Syndrome; Hypertension; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to understand how bariatric surgery affects patients with metabolic syndrome over both the short and long term. We will track changes in blood pressure and other health indicators for up to 10 years after surgery. The goal is to see whether surgery can provide lasting benefits for controlling blood pressure and improving overall health in patients with metabolic syndrome.

DETAILED DESCRIPTION:
Metabolic syndrome (MetS) is a combination of obesity, high blood pressure, abnormal blood sugar, and lipid disorders. It greatly increases the risk of heart disease, stroke, and type 2 diabetes. In Asian populations, MetS often appears at lower body mass index (BMI) levels than in Western countries, making it a growing public health concern even among individuals without severe obesity.

Bariatric surgery has been proven to help patients lose weight and improve blood sugar, blood pressure, and cholesterol levels. However, most studies have been done in patients with severe obesity. There is limited real-world evidence on how surgery affects patients with MetS at lower BMI levels, especially over the long term. In addition, the short-term biological changes that occur immediately after surgery are not fully understood.

This study is a multicenter prospective cohort including patients who had bariatric surgery in three hospitals in China. Patients are being followed for up to 10 years after surgery.

* Early phase: From postoperative day 1 to 7, changes in blood pressure, glucose, and electrolytes are monitored to capture immediate metabolic effects.
* Long-term phase: Follow-up at 3 months, 6 months, 1 year, 5 years, and 10 years is used to assess sustained improvements in weight, blood pressure, glucose, and lipid profiles.

The primary outcome is improvement or resolution of MetS, defined by standardized criteria including BMI, blood pressure, fasting glucose, and lipid levels. Secondary outcomes include changes in individual risk factors, reduction in medication use, and the proportion of patients free of MetS over time.

By providing both short-term and long-term data, this study will clarify how bariatric surgery affects the full course of MetS. The results will help identify patients who may benefit most, guide treatment recommendations, and support better prevention of cardiovascular and metabolic diseases in Asian populations.

ELIGIBILITY:
Inclusion Criteria:

* (1) aged 18-65 years; (2) scheduled to undergo bariatric surgery, including laparoscopic Roux-en-Y gastric bypass (LRYGB) or laparoscopic sleeve gastrectomy (LSG); and (3) met the guideline-based indications for surgery at the time of operation.

Exclusion Criteria:

* (1) coexisting cardiac insufficiency or renal dysfunction; (2) contraindications to bariatric surgery or anesthesia; and (3) refusal to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 65 years who were scheduled to undergo bariatric surgery, including laparoscopic Roux-en-Y gastric bypass (LRYGB) or laparoscopic sleeve gastrectomy (LSG), at three participating medical centers in China. Patients were selected based on guideline-based indications for bariatric surgery at the time of recruitment. For the primary analysis, only patients with hypertension were included, defined as meeting at least one of the following criteria: (1) systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg; (2) self-reported or physician-diagnosed hypertension; or (3) current use of antihypertensive medications. Patients with coexisting cardiac insufficiency, renal dysfunction, contraindications to surgery or anesthesia, or who declined participation were excluded. Additional exclusions during the data analysis phase included patients who experienced severe postoperative adverse events within 7 days, had fewer tha
Sampling Method: Non-Probability Sample
Enrollment: 1581 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Weight | postoperative day 1 to 7, 3 months, 6 months, 1 year, 5 years, and 10 years
Body Mass Index | postoperative day 1 to 7, 3 months, 6 months, 1 year, 5 years, and 10 years
Systolic blood pressure | postoperative day 1 to 7, 3 months, 6 months, 1 year, 5 years, and 10 years
Diastolic blood pressure | postoperative day 1 to 7, 3 months, 6 months, 1 year, 5 years, and 10 years
Status of hypertension | postoperative day 1 to 7, 3 months, 6 months, 1 year, 5 years, and 10 years
Fasting blood glucose | postoperative day 1 to 7, 3 months, 6 months, 1 year, 5 years, and 10 years
Total cholesterol | postoperative day 1 to 7, 3 months, 6 months, 1 year, 5 years, and 10 years
Triglycerides | postoperative day 1 to 7, 3 months, 6 months, 1 year, 5 years, and 10 years

SECONDARY OUTCOMES:
Glycated hemoglobin | postoperative day 1 to 7, 3 months, 6 months, 1 year, 5 years, and 10 years
Low-density lipoprotein (LDL) | postoperative day 1 to 7, 3 months, 6 months, 1 year, 5 years, and 10 years
High-density lipoprotein (HDL) | postoperative day 1 to 7, 3 months, 6 months, 1 year, 5 years, and 10 years
excess weight loss (EWL%) | postoperative day 1 to 7, 3 months, 6 months, 1 year, 5 years, and 10 years
Fasting insulin | postoperative day 1 to 7, 3 months, 6 months, 1 year, 5 years, and 10 years

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Jinshazhou Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - The third xiangya hospital of Central South University, Changsha, Hunan